CLINICAL TRIAL: NCT03432845
Title: Rates and Severity of Postoperative and Post-discharge Nausea and Vomiting of Patients Receiving Sugammadex Versus Neostigmine and Glycopyrrolate for Neuromuscular Block Reversal in Patients Receiving Gastric Bypass Bariatric Surgery
Brief Title: Rates and Severity of PONV for Neuromuscular Block Reversal in Patients Receiving Gastric Bypass Bariatric Surgery
Status: Withdrawn | Type: Observational
Why Stopped: PI left institution
Sponsor: WellSpan Health (Other)
Responsible Party: Principal Investigator, Tara L. Moore, Principal investigator, WellSpan Health
Other Study IDs: IRBNet #1187621-1
Record Dates: First submitted 2018-02-06; First posted 2018-02-14 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sugammadex reversal group: Surgical patients will have their muscle relaxant reversed with sugammadex
  Interventions: Other: compare reversal agents
- Glycopyrrolate / Neostigmine reversal group: Surgical patients will have their muscle relaxant reversed with glycopyrrolate and neostigmine
  Interventions: Other: compare reversal agents

INTERVENTIONS:
Other: compare reversal agents — compare effect of two different approved reversal agents on postoperative and post-discharge nausea and vomiting

SUMMARY:
Patients who require bariatric surgery frequently bring a panoply of pre-existing comorbidities to the operating theatre. With body mass indices routinely in the 50s and 60s, patients who have bariatric surgery frequently have postoperative and post-discharge nausea and vomiting (PONV and PDNV)

DETAILED DESCRIPTION:
There are many causes of post-operative nausea and vomiting in bariatric patients. These include (but are not limited to) the following: 1) mechanical manipulation of the stomach and bowel, 2) post-surgical inflammation of the tissue just operated on, 3) vagal stimulation of the viscera, 4) the administration of volatile anesthetics, 5) the administration of narcotics, 6) the underlying propensity of patient's for post-operative nausea and vomiting, based on prior history, gender, and other factors and 7) the administration of a cholinergic medication for muscle relaxant reversal. From previous work, it is known that alternate techniques are available to mitigate factors two through four, and patient screening has been available to help us determine the likelihood of patients becoming nauseous or vomiting postoperatively (factor #5). However, until the advent of sugammadex, there has been no alternative to factor 6. The use of sugammadex as a reversal agent could dramatically lower the incidence of PONV, while simultaneously providing an excellent level of reversal of neuromuscular blockade. There have been no published studies that have described laparoscopic gastric bypass, sleeve gastrectomy or duodenal switch procedures where complete prevention of PONV has been the result. A secondary objective will be the comparison of pulmonary function before and after surgery between the same two groups. In patients having gastric bypass surgery, not only does PONV aggressively aggravate the tissues which were just surgically manipulated, it also increases the likelihood of decreased ventilatory response, placing patients at risk for aspiration, atelectasis, pneumonia and respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* • > 18 to <= 70 years of age

  * Severe obesity requiring bariatric surgery
  * Willing and able to give informed consent, or if appropriate, have a legally authorized representative capable of giving consent on the participant's behalf
  * Willing to perform the FVC breathing test
  * Willing to be contacted at home via phone

Exclusion Criteria:

* • <18 or >=70 years of age

  * No pregnant patients will be enrolled
  * Patients with documented allergies to anesthesia agents or histories of malignant hyperthermia will not be enrolled.
  * Participants must be eligible to receive elective bariatric surgery
  * Participants who are discharged to skilled care facilities rather than home will not be considered for participation
  * Lacking capacity to provide informed consent
  * Prisoner

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for planned bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
PACU PONV rate and severity | Day of surgery
  The PONV intensity scale measures occurrence and severity. Scoring: Question 1. Have you vomited or had dry retching? A) NO: 0 points, B) Once or Twice: 2 points, C) Three or more times, 50 points. Question 2. Have you experienced a feeling of nausea? If yes, has your feeling of nausea interfered with ADLs, such as being able to get out of bed, being able to move about freely in bed, being able to walk normally, or eating and drinking? A) No: 0 points, B) Sometimes:1 point, C) Often: 2 points, D) All of the time:25 points. Question 3: Has your nausea been mostly: a) Varying? 1 point, b)Constant? 2 points. Question 4: What was the duration of your feeling of nausea (in hours [whole or fraction])? Scoring: Select the highest score of question 1 or 2, then multiply x Q3 x Q4. Minimum 0 points. Maximum score (4 hours) 400 points. Source: Wengritzky R, Mettho T, Myles PS, Burke J, and Kakos A. (2010). BJA, 104 (2), 158-166.

CONTACTS AND LOCATIONS:
Overall Officials: Rich Haas, PhD, Principal Investigator — Principal Investigator

REFERENCES:
- [Background] Dzwonczyk R, Weaver TE, Puente EG, Bergese SD. Postoperative nausea and vomiting prophylaxis from an economic point of view. Am J Ther. 2012 Jan;19(1):11-5. doi: 10.1097/MJT.0b013e3181e7a512. PMID 20634672
- [Background] Hambridge K. Assessing the risk of post-operative nausea and vomiting. Nurs Stand. 2013 Jan 2-8;27(18):35-43. doi: 10.7748/ns2013.01.27.18.35.c9486. PMID 23431652
- [Background] Ziemann-Gimmel P, Goldfarb AA, Koppman J, Marema RT. Opioid-free total intravenous anaesthesia reduces postoperative nausea and vomiting in bariatric surgery beyond triple prophylaxis. Br J Anaesth. 2014 May;112(5):906-11. doi: 10.1093/bja/aet551. Epub 2014 Feb 18. PMID 24554545
- [Background] Wengritzky R, Mettho T, Myles PS, Burke J, Kakos A. Development and validation of a postoperative nausea and vomiting intensity scale. Br J Anaesth. 2010 Feb;104(2):158-66. doi: 10.1093/bja/aep370. Epub 2009 Dec 26. PMID 20037151
- [Background] Gornall BF, Myles PS, Smith CL, Burke JA, Leslie K, Pereira MJ, Bost JE, Kluivers KB, Nilsson UG, Tanaka Y, Forbes A. Measurement of quality of recovery using the QoR-40: a quantitative systematic review. Br J Anaesth. 2013 Aug;111(2):161-9. doi: 10.1093/bja/aet014. Epub 2013 Mar 6. PMID 23471753
- [Background] Myles PS, Wengritzky R. Simplified postoperative nausea and vomiting impact scale for audit and post-discharge review. Br J Anaesth. 2012 Mar;108(3):423-9. doi: 10.1093/bja/aer505. Epub 2012 Jan 29. PMID 22290456
- [Background] Griffith PS, Birch DW, Sharma AM, Karmali S. Managing complications associated with laparoscopic Roux-en-Y gastric bypass for morbid obesity. Can J Surg. 2012 Oct;55(5):329-36. doi: 10.1503/cjs.002011. PMID 22854113
- [Background] Smith, C.A., Haas, R.E., Zepp, J.C. and Klein M., 2016. Improving the quality of post-anesthesia care: An evidence based initiative to decrease the incidence of post-operative nausea and vomiting in the post-anesthesia care unit. Perioperative Care and Operating Room Management, 4, pp. 12-16.
- [Background] Smith C.A., Haas R.E. 2017 Sustaining reductions in postoperative nausea and vomiting after evidence-based practice initiative: A success story. Journal of Health and Social Sciences, 2(2), pp. 149-160.
- [Background] G Power Version 3.0. 10, Faul, F. (2008), Universitat Kiel, Germany
- [Background] Lien, CA and Eikermann, M. Neuromuscular Blockers and Reversal Drugs. Pharmacology and Physiology for Anesthesia, Chapter 19, Saunders, Philadelphia. pp. 325-348.
- [Background] Sheskin, D.J. Handbook of Parametric and Nonparametric Statistical Procedures. CRC Press (1997), Boca Raton.